CLINICAL TRIAL: NCT06582680
Title: Aging, Beta Blockers, and Thermoregulatory Responses
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Crandall, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STU-2024-0644
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Heat Stress; Aging
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: We will first collect participant demographics, medical history, anthropometrics (body mass, height and composition). Individuals will be exposed to 3 hours in a hot environmental condition after receiving the placebo, propranolol, or metoprolol.
  Prior to entering the environmental chamber, baseline data will be collected while resting in a thermoneutral environment. Drug or placebo will be administered. Participants will then enter the environmental chamber and will be seated in a semi-recumbent position on a chair with breathable fabric to minimize impediments to heat dissipation. Periodically throughout the simulated heat-wave participants will lightly exercise to simulate metabolic heat production associated with activities of daily living (~3 metabolic equivalents; METS). Throughout the heat-wave simulation trials we comprehensively evaluate the thermoregulatory and cardiovascular responses.
Who Masked: Participant, Investigator
Masking Description: Neither the participants nor the researchers will know whether the participant received the placebo or one of the beta blocking drugs. Masking will be performed by the research nurse who will know which drug the participant received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Placebo, then Propranolol, then Metoprolol (Experimental)
  Interventions: Other: Ambient Heat
- Placebo, then Metoprolol, then Propranolol (Experimental)
  Interventions: Other: Ambient Heat
- Propranolol, then Placebo, then Metoprolol (Experimental)
  Interventions: Other: Ambient Heat
- Propranolol, then Metoprolol, then Placebo (Experimental)
  Interventions: Other: Ambient Heat
- Metoprolol, then Placebo, then Propranolol (Experimental)
  Interventions: Other: Ambient Heat
- Metoprolol, then Propranolol, then Placebo (Experimental)
  Interventions: Other: Ambient Heat

INTERVENTIONS:
Other: Ambient Heat — Subjects will spend 3-hours in a heat chamber at 41°C and 40% humidity.

SUMMARY:
This study will test the hypothesis that the drugs propranolol and metoprolol will result in greater increases in core body temperature during 3 hours of extreme heat exposure in older adults.

DETAILED DESCRIPTION:
Older individuals are more likely to die or become ill during heat waves. During the 1995 Chicago heat wave, there was 35% increase in hospital admissions for individuals older than 65 years of age. Moreover, adults over the age of 65 have a heat-related death rate that is more than double any other age group. Therefore, with an increasing elderly population that is expected to rise by 60% (to 78 million) by 2035, the causes of this excess mortality must be understood to better protect the ageing United States population. It is notable that selective and non-selective beta blocker drugs are commonly prescribed to older individuals with cardiovascular diseases. In younger individuals exposed to a heat stress, beta blocker administration reduced whole-body sweat rate and skin blood flow responses resulting in greater increases in core body temperature. Notably, nothing is known regarding the effects of beta blockers on thermoregulatory responses during heat exposure in older individuals.

This project will evaluate core body temperature responses to selective and non-selective beta blocker drugs during simulated heat wave exposure in older individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and free of any significant medical problems
* Normal resting electrocardiogram
* 65+ years of age
* Controlled cholesterol of less than 200 mg/dl
* Controlled blood pressure of less than 140/90 mmHg

Exclusion Criteria:

* Known diseases or other chronic conditions requiring regular medical therapy including cancer, diabetes, neurological diseases, uncontrolled hypertension, and uncontrolled hypercholesterolemia
* Serious abnormalities detected on routine screening
* Taking prescribed medications or over-the-counter medications that have known influences on either cardiac function or sweating
* Current smokers, as well as individuals who regularly smoked within the past 3 years
* body mass index ≥31 kg/m2

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Internal temperature | Continuously throughout the 3-hour heat exposure.
  The change in internal temperature to the 3-hour heat exposure will be measured.
Whole body sweat rate | Nude body mass will be measured before and after the 3-hour heat exposure.
  Whole body sweat rate will be measured via changes in pre/post nude body mass.

SECONDARY OUTCOMES:
Heart rate | Continuously throughout the 3-hour heat exposure.
  Heart rate will be measured via electrocardiogram.
Arterial blood pressure | Continuously throughout the 3-hour heat exposure.
  Systolic and diastolic arterial blood pressures will be measured via a brachial blood pressure cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Crandall, PhD, Principal Investigator — Univ of Texas Southwestern Med Ctr
Locations (1):
- IEEM Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No